CLINICAL TRIAL: NCT05935163
Title: Immediate Effects of Bowen Technique Versus Dynamic Soft Tissue Mobilization on Hamstrings Tightness in Chronic Non-specific Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/10
Record Dates: First submitted 2023-05-22; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Hamstring Tightness
Keywords: Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Coventional treatment with Bowen Therapy) (Experimental): Group A will be treated with Bowen Technique in addition to conventional treatment. One session, 45 minutes for technique along with conventional treatment will be given. Technique will be performed for 10 minutes on each limb. The data will be collected at baseline and at 4th week. Follow up will be performed for 4 weeks and 3 sessions will be given each week.
  Interventions: Procedure: Conventional therapy for hamstring tightness; Procedure: Bowen Technique
- Group B (Conventional treatment with DSTM) (Active Comparator): Group B will be treated with Dynamic Soft Tissue Mobilizations (DSTM) in addition to conventional treatment. One session, 45 minutes for technique along with conventional treatment will be given. Technique will be performed for 10 minutes on each limb. The data will be collected at baseline and at 4th week. Follow up will be performed for 4 weeks and 3 sessions will be given each week.
  Interventions: Procedure: Conventional therapy for hamstring tightness; Procedure: Dynamic Soft Tissue Mobilization (DSTM):

INTERVENTIONS:
Procedure: Conventional therapy for hamstring tightness — Conventional Physical therapy will include TENS , hot pack , Hamstring self stretch , Calf self stretching , bridging exercise , piriformis stretch , prone on hands and prone on elbows.
Procedure: Bowen Technique — Bowen Technique:
  1. The patient will assume a full prone-lying position on the plinth.
  2. Sequence of short gentle moves will be applied over hamstrings. Firstly, the thumbs will be placed on top of the hamstrings muscle and the tightness is assessed.
  3. Then, the muscle will be hooked by the thumbs from its lateral edge. Then, gentle pressure will be applied to the point of resistance to challenge the muscle in medial direction, as the thumbs will be flattened in medial direction, the muscle will pluck under the thumbs.
  4. First with the thumbs, then will be followed by the fingers. Often, the hands are placed with a distance of inch of space between the thumbs and fingers so that the hands performed the technique on the muscle easily.
  5. The whole procedure will be repeated again. The treatment time for each session will be 20 minutes for each side.
  Arms: Group A (Coventional treatment with Bowen Therapy)
Procedure: Dynamic Soft Tissue Mobilization (DSTM): — 1. To access the hamstring muscle group, the subject will be asked to attain prone position and deep longitudinal strokes will be applied to the entire muscle group. Once the specific area of hamstring muscle tightness will be located, the remaining treatment will be limited to this target area.
  2. To execute the dynamic intervention, the subject will be requested to move in the supine position with the hip and knee flexed to 90 degree.
  3. Deep longitudinal strokes will be applied in a distal to proximal direction to the area of hamstring tightness and the leg will be passively moved to knee extension. Five strokes will be applied and 20 seconds of shaking is performed at the completion of this technique.
  4. This treatment will be given for 20 minutes on each side.
  Arms: Group B (Conventional treatment with DSTM)

SUMMARY:
Low back pain (LBP) is leading cause of disability and its burden is growing worldwide with an increasing and ageing of population. Poor flexibility or tightness of hamstring muscle has been associated with low back pain. It is a prominent cause of activity limitations and work absenteeism throughout world. Hence this study was designed to find out superior form of effective technique on active knee extension and experience of pain and disability in chronic nonspecific low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is leading cause of disability and it is most leading cause of work absenteeism throughout world. Poor flexibility or tightness of hamstring muscle has been associated with low back pain. Hence this study was designed to find out superior form of effective technique on hamstrings tightness and experience of pain and disability in chronic nonspecific low back pain. This study will also assist to set the foundation for further more studies designing magnificent protocols of treatment for affected population.

ELIGIBILITY:
Inclusion Criteria:

* The patients aged 18-45 years will be included in the study.
* Patients with chronic low back pain (more than 3 months) will be included.
* Both genders.
* 20 to 40 degrees active knee extension loss with hip in 90 degree flexion
* Pain Intensity (moderate to severe) NPRS (4-6 intensity)

Exclusion Criteria:

* Individuals who were receiving treatment for their pain with another(medical treatment) at the same time
* Patients who had undergone vertebral column surgery (less than three months before the time of this study).
* Patients with the infection, neoplasms, metastasis, rheumatoid arthritis, fractures or inflammatory processes were excluded.
* Dislocations of lower limb
* Hypermobility of lower limb joint
* Hamstrings injuries
* Nerve lesions of lower limb

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Active knee extension test | 4 weeks
  active knee extension test, the participant will be in supine-lying position on the treatment bed. Then, participant will flex the hip to 90° while keeping the contralateral hip and knee extended on plinth. The goniometer's fulcrum will be placed on the lateral condyle of the femur at knee joint. The proximal arm of goniometer placed along with the long axis of femur, while moveable arm aligned in line with lateral malleolus. The subject will then extend the knee actively without any pain and tilting of pelvis.
Active straight leg raise (aSLR) | 4 weeks
  The active straight leg raise will be conducted bilaterally three times, and best out of 3 attempts will be recorded. The classic straight leg raise is a complete active test. Each leg is tested individually. When performing the aSLR test, the patient is positioned in supine without a pillow under his/her head. The starting position is described with a distance of 20cm between feet. The patient must rise the leg 20cm from the starting position maintaining the knee in complete extension. The participant will be then asked to rate the difficulty of the task using a 6- point Likert scale. 6-point Likert scale (0= not difficult at all, 1 = minimally difficult, 2 = somewhat difficult, 3= fairly difficult, 4= very difficult, and 5= unable to perform). The test is considered positive when the subjective feeling of fatigue is >3.
The sit-and-reach (SR) tests | 4 weeks
  The subjects sat on the flat surface with their head, back, and hips against a wall, knees straight, legs together, and soles of the feet positioned flat against Sit and Reach box. In keeping this position, the subject will be requested to extend the arms with palms down and lightly touch the index fingers together. The finger-to-box distance will be measured as the distance between the fingertips and the point at which the feet contacted to the box. Then, the subjects will be asked to bend forward slowly and reached as far forward as possible while keeping the knees extended and sliding their hands along a measuring scale placed on the box. Throughout the test, examiner will check to ensure that the heels remained at the box and that the knees are fully extended. The 0 cm mark of the measuring scale represent the position of the feet against the box, with larger values for better performance having higher flexibility.

SECONDARY OUTCOMES:
Pain intensity | 4 Weeks
  Pain status of patients will be assessed using NPRS.
Disability | 4 Weeks
  Disability will be assessed using RMDQ.

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital Department of Rehabilitation, Rawalpindi, Punjab Province, Pakistan